CLINICAL TRIAL: NCT04768946
Title: Using Virtual Technologies to Prevent Injuries in Adolescents With Acquired Brain Injury (ABI)
Brief Title: Using Virtual Technologies to Prevent Injuries in Adolescents With Acquired Brain Injury
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Amy Darragh, Associate Professor, Ohio State University
Other Study IDs: GRT00059789
Record Dates: First submitted 2021-02-10; First posted 2021-02-24 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Acquired Brain Injury; Traumatic Brain Injury; Stroke
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adolescents with Acquired Brain Injury: Adolescents with traumatic brain injury, stroke, and other acquired brain injury ages 12 - 17 will participate in interviews about home safety. They also will have the opportunity to look at and, if desired, try the virtual simulation training system and provide feedback about how to make it more appropriate for adolescents with brain injury, including gamifying it and ensuring appropriate hazards.
- Caregivers of Adolescents with Acquired Brain Injury: Caregivers of adolescents with traumatic brain injury, stroke, and other acquired brain injury will participate in interviews about home safety. They also will have the opportunity to look at the virtual simulation training system and provide feedback about how to make it more appropriate for adolescents with brain injury, including gamifying it and ensuring appropriate hazards.
- Healthcare Workers: This cohort includes health professionals involved in discharge planning and community re-integration of adolescents with ABI. Healthcare workers will participate in interviews about home safety. They also will have the opportunity to look at the virtual simulation training system and provide feedback about how to make it more appropriate for adolescents with brain injury, including gamifying it and ensuring appropriate hazards.

SUMMARY:
The objective of this study is to identify home safety hazards for adolescents with acquired brain injury and to identify adaptations to the home healthcare virtual simulation training system (HH-VSTS) to improve the user experience for adolescents with ABI

DETAILED DESCRIPTION:
This study will determine the home safety hazards that place adolescents with ABI at risk of injury. In addition, the study will determine ways to adapt our current home safety virtual simulation training system, a game based training and assessment that trains home healthcare workers to identify and respond to hazards they encounter in client homes. The study will include interviews with three stakeholders groups: adolescents with ABI, parents of adolescents with ABI, and healthcare providers working with adolescents with ABI to identify home safety hazards encountered by adolescents with ABI. We will demonstrate proof of concept for adolescents with ABI through assessment of safety concerns from multiple perspectives and evaluation of design considerations from our intended user-group. Further, we are applying the HH-VSTS in a novel way to solve an understudied problem in adolescents with ABI. In addition, we will apply a user-centered, participatory approach to assess the design consideration of virtual gaming technologies to health and safety training adolescents with ABI.

ELIGIBILITY:
Inclusion Criteria:

1. adolescent with an acquired brain injury between the ages of 12 - 17 (TBI diagnosis per medical record or self-report for those recruited via word of mouth or community) OR
2. parent/caregiver (18+ years of age) of an adolescent with an acquired brain injury OR
3. a health professional involved in discharge planning and community re-integration of adolescents with an acquired brain injury.
4. For online interview, must have access to a computer or smart tablet with reliable internet access, a microphone, a video camera, and speakers, headphones
5. Speak and read English
6. Able to answer interviewer questions

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will include adolescents with an acquired brain injury between the ages of 12 - 17, parents/caregivers of adolescents with an acquired brain injury, and a health professional involved in discharge planning and community re-integration of adolescents with an acquired brain injury.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Interview Questions | Baseline
  Questions focus on hazard identification, injury risk, factors associated with injury risk.
Usefulness, Usability, and Desirability Assessment | Baseline
  Used to fully assess the usability and appeal of the HH-VSTS, and understand potential modifications
Hazard Rating Scale | Baseline
  Hazards are categorized by frequency of exposure and severity on a two-axis grid, based on participant perceptions.

SECONDARY OUTCOMES:
Interview | one time administration
  Interview questions about safety concerns and perceptions of risk regarding home environment and activity performance

CONTACTS AND LOCATIONS:
Overall Officials: Amy Darragh, PhD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with other researchers secondary to qualitative nature of the data.

REFERENCES:
- [Derived] Anderson SE, Schroedle S, Stamper T, Lundine JP, Patterson ES, DiGiovine CP, Swearingen S, Wengerd LR, Darragh AR. 'I just don't want them to be my patient again': an exploratory mixed-methods study examining provider home safety concerns for adolescents with acquired brain injuries in the US Midwest. Inj Prev. 2024 Nov 11:ip-2024-045326. doi: 10.1136/ip-2024-045326. Online ahead of print. PMID 39532313